CLINICAL TRIAL: NCT06374849
Title: Intraoperative Sufentanil and Chronic Postsurgical Pain in Non-major Scheduled Abdominal Surgery
Acronym: ISPAIN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2023_843_0173
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Postsurgical Pain; Chronic Pain; Abdominal Surgery; Sufentanil; Risk Factors
Keywords: Chronic Postsurgical Pain; Chronic pain; Abdominal surgery; Sufentanil; Risk factors
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone interview — Patient's phone interview 3 months after operating room discharge. The interview consisting of 3 questionnaires to detect the presence of CPSP, its intensity, its characteristics and its related analgesic consumption.

SUMMARY:
Several risk factors for chronic postoperative pain have been identified. A series of studies have shown that administrating intraoperatively a high dose of Remifentanil is associated with an increased incidence of CPSP. These findings highlight a risk factor for CPSP that the anaesthetist can influence on, but they however remain limited to remifentanil. To this day, no study have attempted to evaluate the existence of such an association between the incidence of CPSP and the intraoperative administration of sufentanil doses. Improved knowledge of the long-term nociceptive impact of intraoperative sufentanil administration would enable better therapeutic adaptation according to each patient's risk.

In the field of CPSP, non-major abdominal surgeries remain poorly studied. This is due to their lower risk of CPSP than other surgeries such as orthopaedic, mammary or thoracic surgery. Nevertheless, they constitute a large number of daily surgical procedures. The estimated incidence of CPSP in non-major abdominal surgery appears in several studies to be between 15 and 20% The aim of this study is to evaluate the correlation between the intraoperative administration of sufentanil doses and the incidence of CPSP at 3 months in patients undergoing non-major scheduled abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Non-major scheduled abdominal surgery.
* Patient will receive Sufentanil intraoperatively for induction and maintenance of general anesthesia
* Written or oral informed consent to participate in the study.

Exclusion Criteria:

* Intraoperative complications that are life-threatening or require the surgical procedure to be discontinued.
* Repeat surgery at the same surgical site in less than 3 months.
* Pregnancy.
* Ambulatory surgery.
* Endoscopic surgery.
* Surgery with loco-regional or perimedullary anesthesia without general anesthesia
* Intraoperative use of an opioid other than Sufentanil.
* Hypersensitivity to sufentanil
* Legally protected patients (under judicial protection, guardianship, curatorship).
* Patients suffering from psychiatric pathologies.
* Patients suffering from neurodegenerative pathologies.
* Patients for whom self-assessment of pain using an numerical rating scale (0-10) is not feasible (language barrier, etc…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of CPSP | at 3 months
  Incidence of CPSP at 3 months after non-major scheduled abdominal surgery

SECONDARY OUTCOMES:
Post-operative pain intensity | at 24 hours
  Post-operative pain intensity assessed by NRS of 11 points at 24 hours after operating room discharge
Post-operative pain intensity | at 48 hours
  Post-operative pain intensity assessed by NRS of 11 points at 48 hours after operating room discharge

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No